CLINICAL TRIAL: NCT01656889
Title: A Phase 3 Randomized, Double Blind, Vehicle Controlled Study Investigating the Safety and Efficacy of HP802-247 in the Treatment of Venous Leg Ulcers
Brief Title: Study Investigating the Safety and Efficacy of HP802-247 in the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Healthpoint (Industry)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802-247-09-029
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Venous Leg Ulcers
Keywords: Venous leg ulcer; ulcer; venous stasis; compression; venous; venous stasis ulcer; vlu
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HP802-247 (Experimental): HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 µL (130 µL, one spray, of each solution) containing 0.5 x 106 cells per mL every 14 days.
  Interventions: Biological: HP-802-247
- Vehicle (Placebo Comparator): Vehicle Control (fibrinogen solution & thrombin solution without cells)
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: HP-802-247 — HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 µL (130 µL, one spray, of each solution) containing 0.5 x 106 cells per mL every 14 days.
  Arms: HP802-247
Biological: Vehicle — (fibrinogen solution & thrombin solution without cells)
  Arms: Vehicle

SUMMARY:
This study is being done to find out if an investigational product called HP802-247 can help people with venous leg ulcers. Investigational means that HP802-247 has not been approved by the U.S. Food and Drug Administration (FDA).

This research is being done to compare the efficacy of HP802-247 plus compression therapy against Vehicle plus compression therapy in achieving complete wound closure over the 12-week treatment period. Vehicle looks the same as HP802-247 but contains no cells.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Age ≥ 18 years and of either sex.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Have a venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area ≥ 2.0 cm2 and ≤ 12.0 cm2
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Arterial supply adequacy confirmed
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone.
* Target ulcer duration ≥ 6 weeks but ≤ 104 weeks (24 months).
* Acceptable state of health and nutrition

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, amphotericin B.
* Prior diagnosis of Systemic Lupus Erythematosus with elevated anti-DNA antibody titers, Buerger's disease (thromboangiitis obliterans), current diagnosis of vasculitis, or current diagnosis of claudication.
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit.
* Refusal of or inability to tolerate compression therapy.
* Therapy of the target ulcer with autologous skin graft, Apligraf™, or Dermagraft™ within 30 days preceding the Screening Visit.
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers).
* Any prior exposure to HP802-247 or its vehicle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Chief Medical Officer; Tommy Lee, MSHS, Study Director — Associate Director Clinical Operations; Robert Kirsner, MD, Principal Investigator — Investigator; William Marston, MD, Principal Investigator — Investigator
Locations (45):
- United States (40):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carlsbad, California
  - Castro Valley, California
  - Fresno, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Stockton, California
  - Sylmar, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Hialeah, Florida
  - Miami, Florida
  - South Miami, Florida
  - Tamarac, Florida
  - Chicago, Illinois
  - Jacksonville, Illinois
  - North Chicago, Illinois
  - Springfield, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Las Vegas, Nevada
  - Emerson, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Tulsa, Oklahoma
  - Dunmore, Pennsylvania
  - Wyomissing, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - St. George, Utah
  - Roanoke, Virginia
  - Tacoma, Washington
- Canada (5):
  - Vancovuer, British Columbia
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Sherbrooke, Quebec

REFERENCES:
- [Derived] Marston WA, Ennis WJ, Lantis JC 2nd, Kirsner RS, Galiano RD, Vanscheidt W, Eming SA, Malka M, Cargill DI, Dickerson JE Jr, Slade HB; HP802-247 Study Group. Baseline factors affecting closure of venous leg ulcers. J Vasc Surg Venous Lymphat Disord. 2017 Nov;5(6):829-835.e1. doi: 10.1016/j.jvsv.2017.06.017. PMID 29037354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 43 sites in the US and 5 in Canada; between August 22, 2012 and April 18, 2014; sites included independent and hospital wound clinics and private practice sites.
Pre-assignment Details: Subjects entered a 2-week run-in; subjects whose wound radius decreased by < 0.349 cm/2weeks and met all other inclusion/exclusion (I/E) criteria were eligible for randomization. After completion of the treatment period, subjects entered a three-month follow up period.
Groups:
- Vehicle: Vehicle Control (fibrinogen solution & thrombin solution without cells)
  Vehicle
Period: Treatment Period, 12 Weeks
Arm/Group | HP802-247 | Vehicle
Started | 222 (Randomized (Met all I/E criteria at completion of run-in)) | 225 (Randomized (Met all I/E criteria at completion of run-in))
Completed | 210 (Completed treatment) | 214 (Completed treatment)
Not Completed | 12 | 11
Not completed — Adverse Event | 10 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Moved out of the area | 0 | 2
Period: Post Treatment Follow-Up, 3 Months
Arm/Group | HP802-247 | Vehicle
Started | 210 | 213
Completed | 206 | 204
Not Completed | 4 | 9
Not completed — Death | 1 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Site Closure | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | HP802-247 | Vehicle | Total
Number analyzed (Participants) | 211 | 210 | 421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 136 | 138 | 274
  >=65 years | 75 | 72 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.8) | 61.0 (12.5) | 60.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 82 | 153
  Male | 140 | 128 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 42 | 78
  Not Hispanic or Latino | 175 | 168 | 343
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 43 | 34 | 77
  White | 160 | 167 | 327
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 13 | 22
  United States | 202 | 197 | 399

OUTCOME MEASURES:

1. Primary Outcome: Compare the Treatment Groups for the Proportion of Subjects With Complete Wound Closure Over the 12-Week Treatment Period From Baseline
Description: For each treatment group the area of each subject's target ulcer was measured on a weekly basis, for up to 12 weeks, using a laser-based wound imaging system in conjunction with software to measure area. Following initial closure subjects returned for four weekly visits to confirm wound closure. Wounds that remained closed for four weeks were classified as confirmed closures; if a wound opened at any of the 4 visits it was not considered to have closed. For subjects who dropped from the study, their remaining visit values were imputed using LOCF; wound status of closed was not imputed.
Time Frame: 12 Weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Analysis was by the Cochrane Mantel Haenszel (CMH) test, adjusted for sites, with significance being at P < 0.05
Measure: Number; unit: participants
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 211 | 210
participants
  Wound Closed | 129 | 126
  Wound Not Closed | 82 | 84
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Test type: Superiority or Other; p = 0.5896, Cochran-Mantel-Haenszel; P-value is based on the chi-squared proportion of wounds closed in each group

2. Secondary Outcome: Compare the Efficacy of the Treatment Groups in Achieving Complete Wound Closure, Based on Time in Days to Closure Over the 12-Week Treatment Period From Baseline.
Description: This key secondary outcome was based on a Cox Proportional Hazard Analysis and a Kaplan-Meier survival analysis.
Time Frame: 12 Weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed using the Cox Proportional hazard procedure, with significance being at P < 0.05 and by the Kaplan-Meier survival procedure
Measure: Median (Full Range); unit: days
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 211 | 210
days | 57.0 [8.0 to 115] | 50.0 [6 to 134]
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Test type: Superiority or Other; p = .3675, Regression, Cox

3. Secondary Outcome: Compare the Treatment Groups for the Percentage of Closed Ulcers at Each Visit of the 12-Week Treatment Period From Baseline
Description: Treatment groups were compared for the proportion of wounds closed at each weekly visit. For subjects who dropped from the study, their remaining visit values were imputed using LOCF.
Time Frame: Weekly, over the 12 week treatment period, or until wound closure, which ever occurred first
Population: as for outcome 1
Measure: Number; unit: percentage of Closed Ulcers
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 211 | 210
percentage of Closed Ulcers
  Baseline | 0 | 0
  Treatment Week 01 | 2.4 | 1.9
  Treatment Week 02 | 5.7 | 9.5
  Treatment Week 03 | 13.3 | 19.5
  Treatment Week 04 | 23.7 | 32.4
  Treatment Week 05 | 31.8 | 38.1
  Treatment Week 06 | 38.9 | 44.3
  Treatment Week 07 | 40.8 | 47.6
  Treatment Week 08 | 46.4 | 52.9
  Treatment Week 09 | 49.3 | 55.2
  Treatment Week 10 | 53.6 | 55.7
  Treatment Week 11 | 57.8 | 60.0
  Treatment Week 12 | 63.0 | 62.4
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Treatment Week 01; Test type: Superiority or Other; p = 0.6426, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: HP802-247 vs Vehicle; Treatment Week 02; Test type: Superiority or Other; p = .3843, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: HP802-247 vs Vehicle; Treatment Week 03; Test type: Superiority or Other; p = 0.2792, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: HP802-247 vs Vehicle; Treatment Week 04; Test type: Superiority or Other; p = 0.1502, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: HP802-247 vs Vehicle; Treatment Week 05; Test type: Superiority or Other; p = 0.3823, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: HP802-247 vs Vehicle; Treatment Week 06; Test type: Superiority or Other; p = 0.5528, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: HP802-247 vs Vehicle; Treatment Week 07; Test type: Superiority or Other; p = .02913, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: HP802-247 vs Vehicle; Treatment Week 08; Test type: Superiority or Other; p = 0.3896, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: HP802-247 vs Vehicle; Treatment Week 09; Test type: Superiority or Other; p = 0.3989, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: HP802-247 vs Vehicle; Treatment Week 10; Test type: Superiority or Other; p = 0.8682, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: HP802-247 vs Vehicle; Treatment Week 11; Test type: Superiority or Other; p = 0.8083, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: HP802-247 vs Vehicle; Treatment Week 12; Test type: Superiority or Other; p = 0.6687, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Subjects With Durable Wound Healing Over the 3 Months Following Complete Wound Closure
Description: Subjects who completed the treatment period with confirmed wound closure were followed in the post-treatment period for a further two months to determine their closed wound status (remained closed/reopened), giving a measure of persistence of wound closure following completion of treatment.
Time Frame: Target ulcer status observed at two and three months following initial ulcer closure.
Population: The 285 subjects (HP802-247: 141/222; Vehicle: 144/225) who completed the treatment period with confirmed wound closure.
  Subjects returning for Visit 1 with confirmed wound closure at end of treatment: 134 HP802-247 and 132 Vehicle.
  Subjects returning for Visit 2 with confirmed wound closure at end of treatment: 132 HP802-247 and 131 Vehicle
Measure: Number; unit: participants
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 134 | 132
participants
  Follow-up Visit 1 (2 months), Wounds Closed | 120 | 114
  Follow-up Visit 1 (2 months), Wounds Reopened | 14 | 18
  Follow-up Visit 2 (3 months), Wounds Closed | 118 | 112
  Follow-up Visit 2 (3 months), Wounds Reopened | 14 | 16

5. Secondary Outcome: Change in Pain Associated With the Target Leg at Each of the 12 Double Blind Treatment Weeks
Description: Target leg pain were measured using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects marked their pain level on a 100 mm horizontal line, with a short vertical line across the scale, 0 denoting no pain and 100mm the maximum pain.
Time Frame: Weekly, over the 12 week treatment period, baseline
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed by an ANCOVA, adjusted for site and baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 210 | 210
units on a scale
  Week 01 | -3.74 (1.22) | -2.19 (1.22)
  Week 02 | -4.18 (1.39) | -4.03 (1.38)
  Week 03 | -6.14 (1.4) | -5.91 (1.39)
  Week 04 | -8.2 (1.42) | -6.71 (1.41)
  Week 05 | -10.6 (1.38) | -8.62 (1.37)
  Week 06 | -11.04 (1.53) | -8.2 (1.52)
  Week 07 | -11.57 (1.54) | -9.77 (1.53)
  Week 08 | -11.18 (1.53) | -10.65 (1.53)
  Week 09 | -12.7 (1.5) | -11.26 (1.49)
  Week 10 | -12.55 (1.52) | -11.2 (1.51)
  Week 11 | -12.35 (1.49) | -11.56 (1.48)
  Week 12 | -12.1 (1.49) | -12.27 (1.48)
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Week 01; Test type: Superiority or Other; p = 0.3601, ANCOVA
Statistical Analysis 2: Comparison: HP802-247 vs Vehicle; Week 02; Test type: Superiority or Other; p = 0.9398, ANCOVA
Statistical Analysis 3: Comparison: HP802-247 vs Vehicle; Week 03; Test type: Superiority or Other; p = 0.905, ANCOVA
Statistical Analysis 4: Comparison: HP802-247 vs Vehicle; Week 04; Test type: Superiority or Other; p = 0.4471, ANCOVA
Statistical Analysis 5: Comparison: HP802-247 vs Vehicle; Week 05; Test type: Superiority or Other; p = 0.3004, ANCOVA
Statistical Analysis 6: Comparison: HP802-247 vs Vehicle; Week 06; Test type: Superiority or Other; p = 0.1815, ANCOVA
Statistical Analysis 7: Comparison: HP802-247 vs Vehicle; Week 07; Test type: Superiority or Other; p = 0.399, ANCOVA
Statistical Analysis 8: Comparison: HP802-247 vs Vehicle; Week 08; Test type: Superiority or Other; p = 0.8027, ANCOVA
Statistical Analysis 9: Comparison: HP802-247 vs Vehicle; Week 09; Test type: Superiority or Other; p = 0.4913, ANCOVA
Statistical Analysis 10: Comparison: HP802-247 vs Vehicle; Week 10; Test type: Superiority or Other; p = 0.5227, ANCOVA
Statistical Analysis 11: Comparison: HP802-247 vs Vehicle; Week 11; Test type: Superiority or Other; p = 0.7032, ANCOVA
Statistical Analysis 12: Comparison: HP802-247 vs Vehicle; Test type: Superiority or Other; p = 0.9366, ANCOVA

6. Secondary Outcome: Change in Target Ulcer Pain
Description: Target ulcer pain were measured using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects marked their pain level on a 100 mm horizontal line, with a short vertical line across the scale, 0 denoting no pain and 100mm the maximum pain.
Time Frame: Weekly, over 12 week treament period, baseline
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 210 | 210
units on a scale
  Week 01 | -5.08 (1.08) | -5.05 (1.08)
  Week 02 | -7.59 (1.25) | -6.95 (1.24)
  Week 03 | -10.32 (1.27) | -9.58 (1.26)
  Week 04 | -12.17 (1.3) | -10.26 (1.29)
  Week 05 | -13.15 (1.23) | -13.17 (1.22)
  Week 06 | -15.56 (1.35) | -13.03 (1.34)
  Week 07 | -15.8 (1.38) | -14.51 (1.37)
  Week 08 | -16.28 (1.38) | -14.81 (1.37)
  Week 09 | -17.16 (1.32) | -15.97 (1.31)
  Week 10 | -17.65 (1.32) | -15.91 (1.31)
  Week 11 | -17.34 (1.33) | -16.47 (1.32)
  Week 12 | -17.18 (1.36) | -16.39 (1.35)
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Week 01; Test type: Superiority or Other; p = 0.9853, ANCOVA
Statistical Analysis 2: Comparison: HP802-247 vs Vehicle; Week 02; Test type: Superiority or Other; p = 0.7083, ANCOVA
Statistical Analysis 3: Comparison: HP802-247 vs Vehicle; Week 03; Test type: Superiority or Other; p = 0.6744, ANCOVA
Statistical Analysis 4: Comparison: HP802-247 vs Vehicle; Test type: Superiority or Other; p = 0.2891, ANCOVA
Statistical Analysis 5: Comparison: HP802-247 vs Vehicle; Week 05; Test type: Superiority or Other; p = 0.9923, ANCOVA
Statistical Analysis 6: Comparison: HP802-247 vs Vehicle; Week 06; Test type: Superiority or Other; p = 0.1775, ANCOVA
Statistical Analysis 7: Comparison: HP802-247 vs Vehicle; Week 07; Test type: Superiority or Other; p = 0.499, ANCOVA
Statistical Analysis 8: Comparison: HP802-247 vs Vehicle; Week 08; Test type: Superiority or Other; p = 0.4423, ANCOVA
Statistical Analysis 9: Comparison: HP802-247 vs Vehicle; Week 09; Test type: Superiority or Other; p = 0.5138, ANCOVA
Statistical Analysis 10: Comparison: HP802-247 vs Vehicle; Week 10; Test type: Superiority or Other; p = 0.3409, ANCOVA
Statistical Analysis 11: Comparison: HP802-247 vs Vehicle; Week 11; Test type: Superiority or Other; p = 0.6358, ANCOVA
Statistical Analysis 12: Comparison: HP802-247 vs Vehicle; Week 12; Test type: Superiority or Other; p = 0.6753, ANCOVA

7. Secondary Outcome: Compare the Efficacy of the Treatment Groups in Achieving Complete Wound Closure, Based on the Median Time (in Days) to Closure Over the 12-Week Treatment Period From Baseline.
Description: This key secondary outcome was based on a Kaplan-Meier survival analysis.
Time Frame: 12 weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed using a Kaplan-Meier Survival Analysis, with significance being at P < 0.05.
Measure: Median (Full Range); unit: days to wound closure
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 211 | 210
days to wound closure | 57.0 [8.0 to 115.0] | 50.0 [6.0 to 134.0]
Statistical Analysis 1: Comparison: HP802-247 vs Vehicle; Test type: Superiority or Other; p < 0.05, Kaplan-Meier Survival analysis

ADVERSE EVENTS:
Time Frame: Up to 19 Weeks or subjects who completed 12 weeks of treatment and the post-treatment follow up. For subjects who had wound closure, collection time included the treatment period and the post-treatment period
Description: All subjects randomized to treatment were questioned about AE and were included in the number of participants assessed for safety. The first assessments at each weekly visit were about changes in general health and concomitant medications and the occurrence of AE. Some AE were only collected with respect to the organ system class.
Arm/Group | HP802-247 | Vehicle
Serious Adverse Events (participants affected / at risk) | 17/222 | 21/225
Other Adverse Events (participants affected / at risk) | 119/222 | 107/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=222) | Vehicle (N=225)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Artrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 4 (4)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep-vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=222) | Vehicle (N=225)
Gastrointestinal Disorders (Gastrointestinal disorders) | 7 (9) | 8 (8)
General disorders and administration site conditions (General disorders) | 14 (15) | 11 (14)
Cellulitis (Infections and infestations) | 8 (8) | 10 (15)
Wound infection (Infections and infestations) | 6 (6) | 7 (8)
Injury, poisoining and procedural complication (Injury, poisoning and procedural complications) | 27 (31) | 22 (24)
Wound complication (Injury, poisoning and procedural complications) | 9 (9) | 13 (14)
Infections and Infestations (Infections and infestations) | 39 (48) | 40 (58)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 9 (10) | 4 (5)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 19 (23) | 18 (23)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 15 (17) | 10 (10)
Nervous System Disorders (Nervous system disorders) | 11 (12) | 8 (9)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 71 (99) | 50 (75)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 42 (53) | 31 (44)
Venous Ulcer Pain (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (5)
Vascular Disorders (Vascular disorders) | 11 (13) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less